CLINICAL TRIAL: NCT04096157
Title: A Phase 1 Crossover Study to Assess the Bioequivalence of Isavuconazole Following a Single Dose of Isavuconazonium Sulfate Intravenous Solution Via Nasogastric Tube Compared to a Single Dose of Oral Capsules Under Fasting Conditions in Healthy Subjects
Brief Title: A Study to Assess Isavuconazole Following a Single Dose of Isavuconazonium Sulfate Intravenous Solution Via Nasogastric (NG) Tube Compared to a Single Dose of Oral Capsules Under Fasting Conditions in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 9766-CL-0112
Record Dates: First submitted 2019-09-18; First posted 2019-09-19 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Healthy Subjects
Keywords: Cresemba; isavuconazonium sulfate; isavuconazole
MeSH Terms: interventions — isavuconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Isavuconazonium sulfate IV solution then capsules (Experimental): Participants will first receive a single dose of isavuconazonium sulfate intravenous (IV) solution via nasogastric (NG) tube (test formulation) under fasting conditions on Day 1 of Period 1. After a washout period of 30 days, the participants then receive a single dose of isavuconazonium sulfate capsules (reference formulation) for oral administration under fasting conditions on Day 1 of Period 2.
  Interventions: Drug: Isavuconazonium sulfate IV; Drug: Isavuconazonium sulfate capsules
- Isavuconazonium sulfate capsules then IV solution (Experimental): Participants will first receive a single dose of isavuconazonium sulfate capsules (reference formulation) for oral administration under fasting conditions on Day 1 of Period 1. After a washout period of 30 days, the participants then receive a single dose of isavuconazonium sulfate intravenous (IV) solution via nasogastric (NG) tube (test formulation) under fasting conditions on Day 1 of Period 2.
  Interventions: Drug: Isavuconazonium sulfate IV; Drug: Isavuconazonium sulfate capsules

INTERVENTIONS:
Drug: Isavuconazonium sulfate IV — Intravenous (IV) via nasogastric (NG) tube
  Other Names: Cresemba
Drug: Isavuconazonium sulfate capsules — Oral
  Other Names: Cresemba

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of isavuconazole following a single dose of isavuconazonium sulfate intravenous (IV) solution via nasogastric (NG) tube (test formulation) compared to a single dose of isavuconazonium sulfate capsules for oral administration (i.e., oral capsules administered to nonintubated participants)(reference formulation). In addition, this study will evaluate the safety and tolerability of isavuconazole and the general pharmacokinetic (PK) parameters of isavuconazole when administered as a single dose of isavuconazonium sulfate IV solution via NG tube (test formulation) and a single dose of isavuconazonium sulfate capsules for oral administration (i.e., oral capsules administered to nonintubated participants) (reference formulation) under fasting conditions in healthy male and female participants.

DETAILED DESCRIPTION:
Eligible participants will participate in 2 treatment periods separated by a washout of at least 30 days between investigational product (IP) administrations in each period. Participants will be randomized to 1 of 2 sequences. Participants will be admitted to the clinical unit on day -1 of each period and will be residential for 5 days/4 nights. Participants will receive a single dose of isavuconazonium sulfate IV solution via NG tube (test formulation) or isavuconazonium sulfate capsules for oral administration (i.e., oral capsules administered to nonintubated participants) (reference formulation) under fasting conditions on day 1 of each period. Participants are to remain semirecumbent and avoid lying on either the left or right side for 4 hours postdose. Correct placement of the NG tube will be confirmed using X-ray radiography. Pharmacokinetic samples will be collected predose on day 1 of each period and at multiple time points postdose. Standard safety and tolerability assessments will be conducted. Participants will be discharged from the clinical unit on day 4 of each period on the condition that all required assessments have been performed and that there are no medical reasons for a longer stay in the clinical unit. Participants will return for ambulatory visits to collect pharmacokinetic samples on days 8, 11, 15 and 21 of each period.

The study will be completed with an end-of-study visit (ESV). The ESV will take place 5 to 9 days after day 21 of period 2 or at early discontinuation from the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) range of 18.5 to 32.0 kg/m^2, inclusive and weighs at least 50 kg at screening.
* Female subject is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 30 days after final investigational product (IP) administration.
* Female subject must agree not to breastfeed starting at screening, throughout the study period and for 30 days after final IP administration.
* Female subject must not donate ova starting at first administration of IP, throughout the study period and for 30 days after final IP administration.
* Male subject with female partner(s) of childbearing potential (including breastfeeding partner[s]) must agree to use contraception throughout the treatment period and for 30 days after final IP administration.
* Male subject must not donate sperm during the treatment period and for 30 days after final IP administration.
* Male subject with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy, throughout the study period and for 30 days after final IP administration.
* Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subject has any condition which makes the subject unsuitable for study participation.
* Female subject who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to isavuconazonium sulfate or any components of the formulations used.
* Subject has had previous exposure with isavuconazonium sulfate.
* Subject has any of the liver function tests (alkaline phosphatase [ALP], alanine aminotransferase [ALT], aspartate aminotransferase [AST] and total bilirubin [TBL]) ≥ 1.5 upper limit of normal (ULN) on day -1. In such a case, the assessment may be repeated once.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to first IP administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1.
* Subject has any clinically significant abnormality following the physical examination, ECG (including familial short QT syndrome) and protocol-defined clinical laboratory tests at screening or on day -1.
* Subject has a mean pulse of < 45 or > 90 bpm; mean systolic blood pressure (SBP) >140 mmHg; diastolic blood pressure (DBP) > 90 mmHg (measurements taken in triplicate after the subject has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Subject has a history of peptic or gastric ulcers.
* Subject has a history of sinus disease, sinus allergy, renoplasty or any surgery of the nose, septum or nasal passages or any other abnormality that could impact NG tube placement (e.g., nasal polyps).
* Subject has taken medication or substances via inhalation through the nasal passages within 3 months prior to screening.
* Subject has used any prescribed or nonprescribed drugs (including vitamins and natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to first IP administration, except for occasional use of acetaminophen (up to 2 g/day), topical dermatological products, including corticosteroid products, local anesthetic spray and/or gel (2% Xylocaine) for NG tube placement, hormonal contraceptives and hormone replacement therapy (HRT).
* Subject has smoked, used tobacco-containing products and nicotine or nicotine-containing products (e.g., electronic vapes) within 6 months prior to screening or the subject tests positive for cotinine at screening or on day -1.
* Subject has a history of consuming > 14 units for male subjects or > 7 units for female subjects of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within 2 years prior to screening (note: 1 unit = 12 ounces of beer, 4 ounces of wine, 1 ounce of spirits/hard liquor) or the subject tests positive for alcohol at screening or on day -1.
* Subject has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 or the subject tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) at screening or on day -1.
* Subject has used any inducer of metabolism (e.g., barbiturates and rifampin) in the 3 months prior to day -1.
* Subject has consumed grapefruit, Seville oranges, grapefruit-containing products or Seville orange-containing products within 72 hours prior to day -1.
* Subject has had significant blood loss, donated ≥ 1 unit (450 mL) of whole blood or donated plasma within 7 days prior to day -1 and/or received a transfusion of any blood or blood products within 60 days.
* Subject has a positive serology test for hepatitis A virus antibodies (immunoglobulin M [IgM]), hepatitis B core, hepatitis B surface antigen, hepatitis C virus antibodies or antibodies to human immunodeficiency virus (HIV) type 1 and/or type 2 at screening.
* Subject has abnormal renal function indicated by creatinine above the ULN on day -1. In such a case, the assessment may be repeated once.
* Subject is an employee of Astellas, the study-related contract research organizations (CROs) or the clinical unit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of isavuconazole in plasma: area under the concentration-time curve from the time of dosing extrapolated to time infinity (AUCinf) | Predose on Day 1 and up to Day 21 postdose in each period
  AUCinf will be recorded from the PK plasma samples collected.
PK of isavuconazole in plasma: area under the concentration-time curve from 0 to 72 hours (AUC72) | Predose on Day 1 and up to Day 3 postdose in each period
  AUC72 will be recorded from the PK plasma samples collected.
PK of isavuconazole in plasma: area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast) | Predose on Day 1 and up to Day 21 postdose in each period
  AUClast will be recorded from the PK plasma samples collected.
PK of isavuconazole in plasma: maximum concentration (Cmax) | Predose on Day 1 and up to Day 21 postdose in each period
  Cmax will be recorded from the PK plasma samples collected.

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 61 days
  An AE is any untoward medical occurrence in a participant administered an investigational product (IP), and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of IP whether or not considered related to the IP. An AE is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, hospitalization, or medically important event. Treatment Emergent Adverse Event (TEAE) is defined as any AE which starts, or worsens, after the first dose of study drug through 30 days after the last dose of study drug.
Number of participants with laboratory value abnormalities and/or adverse events | Up to 32 days
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or adverse events | Up to 61 days
  Number of participants with potentially clinically significant vital sign values.
Pharmacokinetics (PK) of isavuconazole in plasma: area under the concentration-time curve extrapolated from time to infinity as a percentage of total AUC (AUCinf(%extrap)) | Predose on Day 1 and up to Day 21 postdose in each period
  (AUCinf(%extrap)) will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of isavuconazole in plasma: apparent clearance (CL/F) | Predose on Day 1 and up to Day 21 postdose in each period
  CL/F will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of isavuconazole in plasma: terminal elimination half-life (t1/2) | Predose on Day 1 and up to Day 21 postdose in each period
  t1/2 will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of isavuconazole in plasma: time of maximum concentration (tmax) | Predose on Day 1 and up to Day 21 postdose in each period
  tmax will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of isavuconazole in plasma: lag time (tlag) | Predose on Day 1 and up to Day 21 postdose in each period
  tlag will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of isavuconazole in plasma: apparent volume of distribution during terminal phase after oral/intravenous administration (Vz/F) | Predose on Day 1 and up to Day 21 postdose in each period
  Vz/F will be recorded from the PK plasma samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Parexel International, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.